CLINICAL TRIAL: NCT07401160
Title: Relationship Between Umbilical Cord Drainage and Postpartum Hemorrhage: A Randomized Single-Blind Clinical Trial.
Brief Title: Umbilical Cord Drainage to Prevent Postpartum Hemorrhage: A Randomized Single-Blind Clinical Trial.
Acronym: CORD-PPH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Autonoma de Honduras (Other)
Responsible Party: Principal Investigator, Ricardo A Gutierrez Ramirez, MD, MSc, FACOG, Ricardo Arturo Gutierrez Ramirez, Universidad Nacional Autonoma de Honduras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PGO-UNAH-49-8-2026
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Postpartum Hemorrhage
Keywords: Cord Drainage; Third Stage of Labor; Obstetric Hemorrhage; Labor Stage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: This is a parallel-group, two-arm, randomized, single-blind trial. Participants are randomly assigned 1:1 to receive either umbilical cord drainage (intervention) or standard active management without drainage (control). Randomization is performed via RedCap. Group assignment is concealed from the outcomes assessors (e.g., personnel measuring blood loss, analyzing lab results, scoring satisfaction scales) to maintain single-blinding and minimize measurement bias, while participants and care providers remain unblinded due to the nature of the procedure.
Who Masked: Outcomes Assessor
Masking Description: The statistician performing the final data analysis will also be blinded to group allocation. Data files for analysis will be coded (Group A, Group B) without identifying the intervention. This additional blinding is implemented to prevent bias during the statistical evaluation of primary and secondary outcomes. All other clinical and research staff involved in patient care, data collection, or immediate postpartum monitoring are unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical Cord Drainage Group (Experimental): Procedure: Umbilical Cord Drainage. Passive drainage of blood from the cut maternal end of the umbilical cord into a calibrated collection drape after birth.
  Interventions: Procedure: Umbilical Cord Drainage
- Standard Care (Control) Group (Sham Comparator): Other: Standard Active Management of Third Stage. Includes administration of uterotonics, controlled cord traction, and monitoring, but no specific cord drainage.
  Interventions: Other: Standard Active Management of Third Stage (No Cord Drainage)

INTERVENTIONS:
Procedure: Umbilical Cord Drainage — Following delivery of the newborn and immediate clamping/cutting of the umbilical cord, the maternal end of the cord is unclamped and allowed to drain passively. The cord is held over a sterile, graduated collection drape (Brass-V Drape) to facilitate the complete, gravity-dependent emptying of the residual placental blood (approximately 50-100 mL) prior to placental delivery. The procedure is completed within 1-3 minutes, after which standard controlled cord traction is applied to assist placental expulsion. This is a non-invasive adjunct to active management of the third stage of labor.
  Arms: Umbilical Cord Drainage Group
Other: Standard Active Management of Third Stage (No Cord Drainage) — This arm receives the standard, evidence-based active management of the third stage of labor, as per institutional protocol, without the specific addition of umbilical cord drainage. The procedure includes immediate administration of a prophylactic uterotonic agent (e.g., oxytocin), delayed cord clamping (as per routine practice), controlled cord traction with counter-pressure on the uterus (Brandt-Andrews maneuver) to assist placental delivery, and uterine massage after placental expulsion. All blood loss is collected and measured in a standard graduated drape. This represents the current standard of care against which the experimental intervention is compared.
  Arms: Standard Care (Control) Group

SUMMARY:
This study aims to analyze whether there is a significant difference in the occurrence of postpartum hemorrhage between women who underwent umbilical cord drainage and those who did not. Variables such as estimated blood loss volume, drop in hemoglobin levels, and the need for additional maneuvers or treatments to control hemorrhage will be examined. The research will be conducted under a parallel-group clinical trial design at the Hospital Escuela Universitario. Post-birth umbilical cord drainage may contribute to a lower frequency of postpartum hemorrhage compared to not performing it.

DETAILED DESCRIPTION:
This is a single-blind, parallel-group, superiority efficacy clinical trial. The intervention involves passive drainage of blood from the umbilical cord immediately after cord clamping and cutting, allowing it to flow into a calibrated drape. The control group receives standard active management of the third stage of labor without cord drainage. The primary objective is to compare postpartum blood loss between the groups. Secondary objectives include comparing pre- and postpartum hemoglobin levels, the need for additional therapeutic interventions (uterotonics, uterine revision, transfusion), incidence of adverse events related to cord management, and maternal satisfaction using the Birth Satisfaction Scale. The study plans to enroll 400 participants (200 per group) over approximately 6 months at a single center.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18-49 years.

Singleton pregnancy.

Gestational age ≥37 weeks.

In active labor with cephalic presentation.

Planned for vaginal delivery.

Capable of providing informed consent.

Exclusion Criteria:

* Planned or emergent cesarean section.

Instrumental delivery (e.g., forceps, vacuum).

Antepartum hemorrhage.

Severe anemia (Hemoglobin <8 g/dL) or specific hematological disorders (e.g., sickle cell disease, thalassemia, hemophilia, thrombocytopenia <100,000/µL).

Use of anticoagulant medication.

Non-cephalic fetal presentation (e.g., breech, transverse).

Refusal to participate or inability to provide informed consent.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only pregnant women
Enrollment: 400 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Postpartum Blood Loss Volume | From delivery until 24 hours postpartum.
  Difference between estimated blood loss volume in the first 24 hours postpartum and an immediate postpartum baseline. Measured using a calibrated drape (Brass-V Drape)

SECONDARY OUTCOMES:
Change in Hemoglobin Levels | Pre-delivery and at 6-24 hours postpartum.
  Difference between pre-delivery and postpartum (6-24 hours) hemoglobin levels (g/dL).
Need for Additional Therapeutic Interventions | First 24 hours postpartum.
  Requirement for additional uterotonics, uterine revision, blood transfusion, or surgical procedures to control hemorrhage.
Incidence of Cord Management-Related Adverse Events | First 24 hours postpartum
  Occurrence of events such as retained placenta, hypovolemic shock.
Maternal Satisfaction Score | At 2 hours postpartum.
  Maternal satisfaction with the intrapartum experience is measured using the validated Birth Satisfaction Scale-Revised (BSS-R). This is a 10-item self-report questionnaire with three subscales: Quality of Care, Women's Personal Attributes, and Stress Experienced During Labor. Items are scored on a 4-point Likert scale (0-3). The total score ranges from 0 to 30, with a higher total score indicating greater birth satisfaction.

CONTACTS AND LOCATIONS:
Locations (2):
- Honduras (2):
  - Hospital Escuela, Tegucigalpa, Francisco Morazán Department
  - Instituto Hondureño de Seguridad Social, Tegucigalpa, Francisco Morazán Department

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make individual participant data (IPD) available. The final decision will depend on the specific requirements of the target publication journal, further consultation with the local ethics committee regarding data sharing agreements, and a thorough assessment of our capacity to properly anonymize the data while preserving its scientific value for secondary analysis.

REFERENCES:
- [Background] Koshkin ES. A review of the genus Dodia Dyar, 1901 (Lepidoptera: Erebidae, Arctiinae) with description of a new remarkable species from the Russian Far East. Zootaxa. 2024 May 27;5458(1):53-72. doi: 10.11646/zootaxa.5458.1.2. PMID 39646951